CLINICAL TRIAL: NCT00319280
Title: Proximal Tibial Open Wedge Osteotomy. Stability and Healing Evaluated in a Clinical Prospective, Randomized Trial Using RSA.
Brief Title: Proximal Tibial Open Wedge Osteotomy. A Clinical Prospective, Randomized RSA-trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Company CCBR A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-01-004-ML
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Osteotomy; Healing; Roentgen Stereometric Analysis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Minced Iliac Crest autograft in osteotomysite
  Interventions: Procedure: bonesubstitution (Calcibon, Iliac Crest Bonegraft, control)
- 2 (Experimental): Injectable calcium phosphate cement in osteotomysite
  Interventions: Procedure: bonesubstitution (Calcibon, Iliac Crest Bonegraft, control)
- 3 (Active Comparator): Local autograft in the osteotomysite serves as control
  Interventions: Procedure: bonesubstitution (Calcibon, Iliac Crest Bonegraft, control)

INTERVENTIONS:
Procedure: bonesubstitution (Calcibon, Iliac Crest Bonegraft, control) — Osteotomysite are filled with Calcibon (an injectable calcium phosphate cement) or Minced Iliac Crest Bonegraft og local graft as control

SUMMARY:
In the treatment of osteoarthritis of the medial compartment of the knee, Open wedge high tibial osteotomy is a good choice of treatment for the young and active patient.

However it leaves an open gap which has to be filled with a bone substitute and requires stable fixation.

Hitherto the golden standard has been autograft taken from iliac crest but there are donorsite related problems and limited amount available.

Recently injectable and resorbable calciumphosphate-cements have been introduced and used with promising results in fractures of the distal radius, calcaneus and lateral tibial condyle.

These new cements seem to be a good alternative to other bone substitutes providing high initial strength that might promote early mobilisation; it resorbs and promotes osteoconduction securing safe healing.

The aim of the present study is to evaluate whether there is any difference in clinical outcome, correction, stability and healing in open-wedge osteotomies with three different bone substitutes: Autograft from iliac crest and the injectable calciumphosphate-cement Calcibon and as control a group with an empty gap.

Osteosynthesis is performed with the Dynafix® system (EBI) The investigation is performed as a randomised prospective clinical trial including 45 patients with a planned 2 years follow-up period.

Clinical outcome is evaluated with: Hospital of special surgery score, KOOS, SF 12 and Lysholm score.

Routine standing x-rays is performed. Stability is assessed with Roentgen Stereophotogrammetric Analysis (RSA) that provides the opportunity of exact 3-dimensional measuring of eventual loss of correction.

This combined with urine and serum bone-healing markers gives a very precise picture of the healing in the bone-gap.

To asses the cartilage of the knee MRI is performed and biochemical markers fore Collagen type II degradation are measured.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of medial compartment of the knee, Ahlbäck gr. 1-2
* Candidate for proximal tibial medial open-wedge osteotomy
* Signed informed consent

Exclusion Criteria:

* Prednisolone treatment.
* NSAID treatment.
* BMI > or = 35.
* Previous surgery in lateral knee compartment.
* Secondary Arthrosis following fracture(s) of the tibial condyle(s).
* Lack of informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Migration in mm measured with RSA (Roentgen Stereometric Analysis) | postoperative, at 3 month, 1 and 2 years

SECONDARY OUTCOMES:
Hip-Knee-Ankle axis | 3 month, 1 and 2 years.
MR of the knee | 4 weeks preoperative, preoperative, at 1 and 2 years postoperative.
Markers of chondral degradation | preoperative, at 6 weeks, 3 month, 1 and 2 years postoperative
Markers of bone synthesis and degradation | preoperative, at 6 weeks, 3 month, 1 and 2 years postoperative
Clinical scores: KOOS, Lysholm, SF12, Knee Score | Preoperatively, Postoperatively, 6 weeks, 3 months, 1 year and 2 years
Histomorphometric evaluation of bone healing and osseous integration of cement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lind-Hansen, MD, Principal Investigator — Northern Orthopaedic Division, Denmark
Locations (1):
- Northern Orthopaedic Division, Klinik Farsoe, Aalborg University Hospital, Farsø, Northern Jutland, Denmark